CLINICAL TRIAL: NCT00732953
Title: Prevention of Restenosis After Genous Stent Implantation Using a Paclitaxel Eluting Balloon in Coronary Arteries - a Randomized Clinical Trial.
Brief Title: Prevention of Restenosis After Genous Stent Implantation Using a Paclitaxel Eluting Balloon in Coronary Arteries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: B. Braun Melsungen AG (Industry); OrbusNeich (Industry)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UULM-JW-GP
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease
Keywords: patients with coronary artery disease; percutaneous coronary intervention; stent implantation; paclitaxel eluting balloon; angiographic follow-up; clinical follow-up
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Genous stent implantation with paclitaxel-eluting balloon therapy
  Interventions: Device: Genous stent implantation with paclitaxel-eluting balloon dilation
- 2 (Active Comparator): Genous stent implantation
  Interventions: Device: Genous stent implantation

INTERVENTIONS:
Device: Genous stent implantation with paclitaxel-eluting balloon dilation — Genous stent implantation with paclitaxel-eluting balloon therapy
  Arms: 1
Device: Genous stent implantation — Genous stent implantation
  Arms: 2

SUMMARY:
Percutaneous coronary intervention with stent implantation is limited on the one hand by restenosis due to smooth muscle cell proliferation and on the other hand by stent thrombosis due to incomplete or not sufficient enough endothelialization of stent struts. The Genous stent implantation allows a rapid layer over the stent struts with endothelial progenitor cells allowing a fast endothelialization and probably reducing the risk of stent thrombosis. Local therapy with drug-eluting balloons administering paclitaxel has been shown to reduce restenosis in in-stent restenosis and de-novo lesions in vessels with small reference diameter. The combination of a paclitaxel-eluting balloon and Genous stent implantation may summarized both advantages: a rapid endothelialization limiting the number of stent thrombosis and on the other hand a reduction of smooth muscle cell proliferation minimizing the risk of restenosis with the subsequent need for revascularization.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old
* lesion in native coronary artery
* de-novo stenosis
* indication for revascularization (angina status, myocardial ischemia, positive stress test, pathologic FFR)
* range of reference diameter 2.5 to 4.0mm

Exclusion Criteria:

* lesion in saphenous vein graft
* chronic total occlusion
* bifurcation lesion requiring stenting of main and side branch
* left main stenosis
* restenosis
* in-Stent restenosis
* contraindication for dual antiplatelet therapy for the following 6 months
* coronary aneurysm in target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Late loss | 6 months

SECONDARY OUTCOMES:
Diameter stenosis | 6 months
Binary restenosis rate | 6 month
Late loss index | 6 months
Target lesion revascularization | 2, 6, 12, 24, 36, 48, 60 months
Target vessel revascularization | 2, 6, 12, 24, 36, 48, 60 months
Major adverse cardiac events | 2, 6, 12, 24, 36, 48, 60 months
Stent thrombosis | 2, 6, 12, 24, 36, 48, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD, Principal Investigator — University of Ulm
Locations (3):
- Germany (3):
  - Klinikum Coburg, Coburg
  - University of Ulm, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen

REFERENCES:
- [Background] Wohrle J, Birkemeyer R, Markovic S, Nguyen TV, Sinha A, Miljak T, Spiess J, Rottbauer W, Rittger H. Prospective randomised trial evaluating a paclitaxel-coated balloon in patients treated with endothelial progenitor cell capturing stents for de novo coronary artery disease. Heart. 2011 Aug;97(16):1338-42. doi: 10.1136/hrt.2011.226563. Epub 2011 May 26. PMID 21617163
- [Derived] Seeger J, Markovic S, Birkemeyer R, Rittger H, Jung W, Brachmann J, Rottbauer W, Wohrle J. Paclitaxel-coated balloon plus bare-metal stent for de-novo coronary artery disease: final 5-year results of a randomized prospective multicenter trial. Coron Artery Dis. 2016 Mar;27(2):84-8. doi: 10.1097/MCA.0000000000000314. PMID 26479969